CLINICAL TRIAL: NCT04250142
Title: Effect of Pulp Protection After Selective Carious Tissue Removal in Permanent Teeth, a Randomized Controlled Clinical Trial
Brief Title: Pulp Protection in Selective Carious Tissue Removal
Acronym: PULPROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Responsible Party: Principal Investigator, Rodrigo A. Giacaman, DDS, PhD, Full Professor, University of Talca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CM-11/2018
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
Keywords: Dental caries; Selective Caries Removal; Self-etching adhesive; Composite Resin; Glass ionomer; Cavity lining; Minimally invasive dentistry; Deep caries lesions
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A double blinded randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will not know the type of treatment they will receive. The data analysis will be carried out assigning a letter to the treatment arms, and the identity of the arms will not be revealed up until the end of the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Glass Ionomer (Active Comparator): Selective removal of carious tissue to soft dentin. Deep carious dentin will be lined by a conventional glass ionomer, followed by a composite resin restoration.
  Interventions: Device: Glass Ionomer
- Self-etching Adhesive (Experimental): Selective removal of carious tissue to soft dentin. Deep carious dentin will not be lined and a self-etching adhesive will cover the tissue, followed by a composite resin restoration.
  Interventions: Device: Self-etching Adhesive

INTERVENTIONS:
Device: Self-etching Adhesive — A Self-etching adhesive will be used to cover deep carious dentin after a selective removal of caries lesion to soft dentin procedure.
  Other Names: Self-conditioning Adhesive; Self-etching primer; Single Bond Universal (3M)
  Arms: Self-etching Adhesive
Device: Glass Ionomer — A conventional glass ionomer will be used to cover deep carious dentin after a selective removal of caries lesion to soft dentin procedure.
  Other Names: Conventional Glass Ionomer; Ketac Molar (3M)
  Arms: Conventional Glass Ionomer

SUMMARY:
Although selective removal of carious tissue to soft dentin (SRCT-S) has been proposed as the standard of care for the management of deep dentin caries, it is unclear whether a cavity liner is necessary. This double blinded randomized controlled clinical trial aims to analyze the behavior of a resin restoration performed after SRCT-S for deep dentin caries, treated either with a Glass Ionomer or only with a Self-Etching Adhesive, in permanent teeth. The study will include 142 restorations allocated to either experimental arm. After 12 and 24 months, restoration survival, pulp response and radiographic lesion progression will be assessed.

DETAILED DESCRIPTION:
Introduction: Minimally invasive dentistry has been proposed as an conceptual framework for the conservative management of caries lesions. This approach allows reducing potential adverse effects derived from the conventional treatment, including the loss of pulp vitality. Complete removal carious tissues compromising deep dentin significantly increases the risk of pulp exposure and post-operative symptoms, leading in many cases, to the need for endodontic treatment, with the subsequent high costs and low coverage for the population. In this context, a new technique for the management of deep caries lesions has been introduced called selective removal of carious tissue to soft dentin (SRCT-S), which partially removes only the outer layer of the affected tissue, leaving carious tissue in the pulpal wall, but not on the lateral walls of the operatory cavity. This procedure has been reported in several studies, with lower clinical time, cheaper cost and lower discomfort for the patient. The SRCT-S aims to preserve pulp vitality, prevent access of nutrients to carious tissue, stopping the caries process and preserving a greater amount of dental structure. Although the SRCT-S technique has proven effective compared to conventional treatments, it is unclear and with insufficient evidence about how to manage the remaining carious tissue and whether a cavity lining agent is needed. This decision may have important clinical implications, but there is no general consensus, strongly suggesting further research. Objective: To analyze the behavior of a resin restoration performed after SRCT-S for deep dentin caries, treated either with a Glass Ionomer or only with a Self-Etching Adhesive, in permanent teeth. Methodology: A double blinded randomized controlled clinical trial was devised. Trained dentists will treat the 142 restorations included in deep dentin carious lesions of permanent molars, at the dental clinics of the University of Talca. After recruiting, patients will be randomly assigned to the experimental groups: Group 1: (n=71) no cavity lining, treating carious tissue with self-conditioning adhesive followed by composite resin restoration and Group 2: (n=71) remaining carious tissue covered with a conventional glass ionomer followed by composite resin restoration. The dependent variables (outcomes) will be; a. clinical: restoration survival and pulp response and b. radiographic: lesion progression. Clinical and radiographic outcomes will be monitored annually at 12 and 24 months. The analysis of the restorations and the pulp response will be performed with Weibull regression. The Friedman test will be applied for the analysis of the data regarding radiographic subtraction, (p≤0.05). Given the lack of studies on the subject with longitudinal evaluations, this project is expected to contribute relevant evidence that impacts the generation of novel guidelines for the management of deep dentin caries. Additionally, the results will contribute evidence to increase the support to a more conservative clinical behavior.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a permanent molar or premolar with a deep caries lesion that compromises from the inner half of the dentin (determined by radiographic examination).
* Tooth restorable by a direct resin restoration.
* Absence of pulp sensibility verified by cold test
* Absence of a history of spontaneous pain or vertical and horizontal percussion.
* Absence of periapical lesion, verified through periapical radiographs.
* Primary injury.

Exclusion Criteria:

* Systemic conditions with poor control or uncompensated.
* Cervical margin of the cavity in dentin or root cement.
* Tooth already restored or with secondary caries.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Restoration integrity | 2 years
  The FDI Criteria will be used for the direct clinical evaluation of restorations.
Pulp vitality | 2 years
  Pulp vitality will be evaluated by means of symptoms reported by the patient, normal response upon thermal tests, no pain upon percussion, absence of periapical lesions (periapical radiography) and absence of infectious processes such as fistula.

SECONDARY OUTCOMES:
Radiographic progression | 2 years
  Lesion progression at the x-ray will be monitored through qualitative analysis with the technique of digital subtraction of the radiographic images (radiolucent area under restorations) over time.
Changes in pulp chamber morphology | 2 years
  For the qualitative analysis of the depth of the lesion and the deposition of tertiary dentin, the pairs of radiographic images (baseline radiographs versus control radiographs) will be assessed and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Muñoz Sandoval, DDS, Study Director — University of Talca
Locations (1):
- Faculty of Health Sciences, Talca, No State, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maltz M, Alves LS, Jardim JJ, Moura Mdos S, de Oliveira EF. Incomplete caries removal in deep lesions: a 10-year prospective study. Am J Dent. 2011 Aug;24(4):211-4. PMID 22016914
- [Background] Maltz M, Koppe B, Jardim JJ, Alves LS, de Paula LM, Yamaguti PM, Almeida JCF, Moura MS, Mestrinho HD. Partial caries removal in deep caries lesions: a 5-year multicenter randomized controlled trial. Clin Oral Investig. 2018 Apr;22(3):1337-1343. doi: 10.1007/s00784-017-2221-0. Epub 2017 Oct 8. PMID 28988345
- [Background] Bjorndal L, Reit C, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Thordrup M, Dige I, Nyvad B, Fransson H, Lager A, Ericson D, Petersson K, Olsson J, Santimano EM, Wennstrom A, Winkel P, Gluud C. Treatment of deep caries lesions in adults: randomized clinical trials comparing stepwise vs. direct complete excavation, and direct pulp capping vs. partial pulpotomy. Eur J Oral Sci. 2010 Jun;118(3):290-7. doi: 10.1111/j.1600-0722.2010.00731.x. PMID 20572864
- [Background] Bjorndal L, Fransson H, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Hedenbjork-Lager A, Dige I, Thordrup M. Randomized Clinical Trials on Deep Carious Lesions: 5-Year Follow-up. J Dent Res. 2017 Jul;96(7):747-753. doi: 10.1177/0022034517702620. Epub 2017 Apr 14. PMID 28410008
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774